CLINICAL TRIAL: NCT01570556
Title: Clinical Impact of Bacteriuria on Chronic Inflammation in Asymptomatic Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 193/11
Record Dates: First submitted 2012-03-15; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Inflammation on Dialysis; Bacteriuria in Hemodialysis Patients
Keywords: Hemodialysis; Inflammation; Bacteriuria; Interleukin 6; C reactive protein
MeSH Terms: conditions — Inflammation; Bacteriuria

ARMS (2):
- Patients with positive culture, treatment group (Active Comparator): These asymptomatic patients with positive urinary culture, seven days of antibiotics will be given according to the bacteriogram sensitivity.
  Interventions: Other: Antibiotic treatment
- Patients with positive culture, observation only (No Intervention): These asymptomatic patients with positive urine culture, will be observed only during the study period.

INTERVENTIONS:
Other: Antibiotic treatment — In patients with positive urinary culture, seven days of antibiotics will be given orally according to the bacteriogram sensitivity.
  Arms: Patients with positive culture, treatment group

SUMMARY:
When considering occult infections during the diagnostic workup of inflammation in Hemodialysis (HD) patients, the urine-deprived bladder is frequently dismissed as potential site of infection. The urinary tract, even in end stage renal disease (ESRD) patients on hemodialysis may represent a significant reservoir for infection. Delayed diagnosis is a relevant issue because the urinary tract is often overlooked as a source of infection in dialysis patients, especially because of absence of urinary tract infection (UTI) symptoms in HD patients. Contributing factors to asymptomatic UTI in HD patients include the presence of low urine volume, bladder stasis, and the fact that UTI symptoms are mostly related to voiding, which is reduced or absent in these patients. Persistence of asymptomatic bacteriuria and UTI may be related to higher levels of inflammatory markers in HD population. In view of the association between cardiovascular disease and cardio-vascular and all-cause mortality with inflammation, as expressed by elevated CRP and/or IL-6 levels in HD patients, the investigators questioned whether presence of asymptomatic UTI could contribute to elevated levels of inflammatory markers in patients with ESRD on maintenance HD therapy. Such a finding would provide a potential link between a treatable infection and a potential cardiovascular risk factor in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18 years, in chronic hemodialysis treatment at least 3 months
2. Stable and adequate hemodialysis treatment three months prior to participation in study as defined by Kt/V > 1.2 and hemodialysis performed at least 3 times weekly
3. Patients with native A-V Fistula or graft
4. Informed consent obtained before any trial-related activities

Exclusion Criteria:

1. Patients with an indwelling catheters
2. Patients with periodontitis
3. Patients with diabetic foot
4. Patients with active malignant disease or liver cirrhosis
5. Patients on chronic treatment with steroids on doses > 10 mg/day Prednisone (or equivalent)
6. Patients treated with immunosuppressive agents
7. Patients suffering from

   * Acute vasculitis
   * Severe systemic infections
   * Heart failure (NYHA class III-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum inflammatory markers (CRP, IL-6) | 3 months, 6 months, and 12 months

SECONDARY OUTCOMES:
Cardio-vascular events | 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department, Assaf Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Background] Beberashvili I, Sinuani I, Azar A, Yasur H, Shapiro G, Feldman L, Averbukh Z, Weissgarten J. IL-6 levels, nutritional status, and mortality in prevalent hemodialysis patients. Clin J Am Soc Nephrol. 2011 Sep;6(9):2253-63. doi: 10.2215/CJN.01770211. Epub 2011 Aug 18. PMID 21852667